CLINICAL TRIAL: NCT02550834
Title: The Effects of Indoors Curling Exercise in Persons With Chronic Spinal Cord Injury on Control Capabilities of Trunk Movements: a Randomized-controlled Trial.
Brief Title: Wheelchair Indoors Curling With SCI patients_RCT
Acronym: SCI-RCT
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: HES-SO Valais-Wallis (Other)
Collaborators: Clinique Romande de Readaptation (Network); Uniklinik Balgrist, Zürich (Unknown)
Responsible Party: Principal Investigator, Mittaz Hager Anne-Gabrielle, Professor, HES-SO Valais-Wallis
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 44408
Record Dates: First submitted 2015-09-09; First posted 2015-09-16 (Estimated); Last update posted 2016-02-24 (Estimated); Status verified 2016-02

CONDITIONS: Spinal Cord Injury
Keywords: Core stability; Indoors curling exercises; Motivation
MeSH Terms: conditions — Spinal Cord Injuries

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Experimental : Curling group (Experimental)
  Interventions: Other: Wheelchair indoors curling training
- Control : Usual care group (No Intervention)

INTERVENTIONS:
Other: Wheelchair indoors curling training — 8x 90 minutes of training and playing indoors curling in 4 weeks
  Arms: Experimental : Curling group

SUMMARY:
This study investigates if, patients with diagnosed chronic spinal cord injury will benefit from an Indoor Curling Exercise program on their control capabilities of trunk movements and on their intrinsic motivation for physical activity. Half of participants will receive 8 training-sessions during 4 weeks, while the other will receive usual care.

DETAILED DESCRIPTION:
Spinal cord injury (SCI) is a catastrophic event that can be devastating and costly in human and social terms. These patients require multidisciplinary and interdisciplinary treatment. Physiotherapy is important factor in SCI rehabilitation.

The objectives of physiotherapists are manifold and include the development of the force of healthy muscles, the teaching of transfer techniques, the maintenance of joint motion and of the body map, and the reestablishment of sitting balance in order for the patients to regain their autonomy.

Maintaining postural stability when seated is a challenge for people with a SCI as their sensory and motor systems in their trunk, lower and upper extremities have been damaged to different degrees. To train this postural stability, physiotherapists include many interventions. Physical activities in sport therapy are some of them. In addition to usual physical activities (basketball, tennis, wheelchair running,…) the investigators propose to practice wheelchair Indoors Curling Exercise with wooden Curling Stones.

ELIGIBILITY:
Inclusion Criteria:

* Traumatic, non-traumatic or ischemic Spinal Cord Injury with complete or incomplete para- or tetraplegia
* Complete spinal cord status (ASIA Score)
* Sitting capabilities ≥ 4 hours
* Capability to bench 20° forward in trunk flexion
* Signed informed consent after being informed

Exclusion Criteria:

* Progressives pathologies
* Problem in vestibular system
* Severely impaired vision
* Tetraplegia without hand function
* Acute pain
* Contraindications on ethical grounds
* Previously reduced capabilities of cooperation
* Know or suspected non-compliance

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2015-08; Primary Completion 2015-12 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
Sitting balance | 8 weeks
  Control capabilities of trunk movement (6-channel inertial sensor by 25 cycles per minute, back-and-forth trunk movements), Modified Functional Reach Test

SECONDARY OUTCOMES:
Intrinsic Motivation | 8 weeks
  Intrinsic Motivation Inventory (IMI)

CONTACTS AND LOCATIONS:
Locations (2):
- Switzerland (2):
  - Uniklink Balgrist, Zurich, Canton of Zurich
  - Clinique romande de réadaptation CRR-SUVA, Sion, Valais